CLINICAL TRIAL: NCT04642820
Title: Drugs Brain and Behavior
Brief Title: Drugs Brain and Behavior (DDP)
Acronym: DDP
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IRB20-0364; R01DA002812 (NIH)
Record Dates: First submitted 2020-11-18; First posted 2020-11-24 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2023-12

CONDITIONS: Stimulant Use
MeSH Terms: interventions — Methamphetamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo Then Methamphetamine (Experimental): Participants first receive placebo at their first session in the laboratory. Then will return to the laboratory 72 hours later and will receive 20 mg methamphetamine.
  Interventions: Drug: Methamphetamine; Drug: placebo oral tablet
- MethamphetamineThen Placebo (Experimental): Participants first receive 20 mg methamphetamine at their first session in the laboratory Then will return to the laboratory 72 hours later and will receive placebo.
  Interventions: Drug: Methamphetamine; Drug: placebo oral tablet

INTERVENTIONS:
Drug: Methamphetamine — Participants will be given 20 mg of Methamphetamine.
Drug: placebo oral tablet — Participants will be given a placebo capsule that will only contain lactose.

SUMMARY:
In this project, we will examine individual differences in the effects of a stimulant drug, methamphetamine (MA), on mesolimbic reward function using fMRI.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 19 and 26
* Right Handed
* Less than 4 alcohol or caffeinated beverages a day.

Exclusion Criteria:

* High blood pressure
* Any medical condition requiring regular medication
* Individuals with a current (within the last year) DSM-IV Axis 1 diagnosis
* Individuals with a history of dependence on stimulant drugs
* Women who are pregnant or trying to become pregnant.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 138 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2024-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harriet de Wit, Principal Investigator — Principal Investigator
Locations (1):
- University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo Then Methamphetamine | MethamphetamineThen Placebo
Started | 69 | 69
Completed | 57 | 56
Not Completed | 12 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Then Methamphetamine | MethamphetamineThen Placebo | Total
Number analyzed (Participants) | 57 | 56 | 113
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.3 (4.3) | 25.3 (3.7) | 24.8 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 28 | 56
  Male | 29 | 28 | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 14 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 32 | 28 | 60
  More than one race | 8 | 1 | 9
  Unknown or Not Reported | 9 | 9 | 18
Region of Enrollment [Number; unit: participants]
  United States | 57 | 56 | 113

OUTCOME MEASURES:

1. Primary Outcome: Change in SUbjective Effects as Assessed by Score on "Feel Drug", "Feel High", "Like Drug", and "Want More" Sub-scales of Drug Effects Questionnaire (DEQ).
Description: Participants will complete The Drug Effects Questionnaire during the initial baseline session to determine their subjective stimulant profile. The Dug Effects Questionnaire (DEQ) is a visual analog scale questionnaire that assesses the extent to which subjects experience four subjective states: "Feel Drug", "Feel High", "Like Drug", and "Want More". All sub-scales are scored on a visual analogue scale (Scroll bar on computer screen) ranging from 0-100. 100 represents the highest score for that subjective state, and the higher the score, the worse the outcome.
Time Frame: Time Frame: Day 1(baseline), 3
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo: placebo oral tablet: Participants will be given a placebo capsule that will only contain lactose.
Arm/Group | Placebo | Methamphetamine
Number analyzed (Participants) | 113 | 113
score on a scale
  DEQ Feel - Change from baseline | 19.2 (21.6) | 57.8 (25.7)
  DEQ Like - Change from baseline | 28.6 (28.0) | 76.3 (26.5)
  DEQ Dislike - Change from baseline | 25.2 (28.7) | 26.8 (25.8)
  DEQ High - Change from baseline | 13.9 (19.4) | 48.7 (29.4)
  DEQ Want more - Change from baseline | 22.3 (28.1) | 69.1 (28.7)
Statistical Analysis 1: Comparison: Placebo vs Methamphetamine; Test type: Superiority; p = .05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 1 month, through study completion
Arm/Group | Placebo Then Methamphetamine | MethamphetamineThen Placebo
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/56
Other Adverse Events (participants affected / at risk) | 0/57 | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-09): https://cdn.clinicaltrials.gov/large-docs/20/NCT04642820/Prot_SAP_000.pdf